CLINICAL TRIAL: NCT00582296
Title: Adherence to Comprehensive, Multi-Organ Screening Recommendations in Patients With Lynch Syndrome
Brief Title: Multi-Organ Screening Recommendations in Patients With Lynch Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 04-144
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Lynch Syndrome
Keywords: Lynch syndrome; 04-144
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: multi-organ follow-up
  Interventions: Behavioral: questionnaires, telephone interview, optional blood drawn
- 2: control follow-up
  Interventions: Behavioral: questionnaires, telephone interview and optional blood drawn

INTERVENTIONS:
Behavioral: questionnaires, telephone interview, optional blood drawn — Initial CGS Visit (All Prospective Participants)Clinical assessment (screening, family & personal history of CA, surgeries) 6 Month Follow-Up Phone Interview (Prospective) Follow-Up Questionnaire (prospective and retrospective) Retrospective Initial Interview Participants may also donate an additional blood, serum, saliva, urine, or stool sample for research, (in addition to the blood drawn for clinical testing) or for the sole purpose of research testing (in absence of clinical testing or prior external testing).
  Groups: 1
Behavioral: questionnaires, telephone interview and optional blood drawn — Initial CGS Visit (All Prospective Participants)Clinical assessment (screening, family & personal history of CA, surgeries) 6 Month Follow-Up Phone Interview (Prospective) Follow-Up Questionnaire (prospective and retrospective) Retrospective Initial Interview Participants may also donate an additional blood, serum, saliva, urine, or stool sample for research, (in addition to the blood drawn for clinical testing) or for the sole purpose of research testing (in absence of clinical testing or prior external testing).
  Groups: 2

SUMMARY:
The purpose of this study is to examine how people with a family history of colon cancer and other related cancers respond to recommendations for cancer screening after genetic counseling. The purpose of your participation would be to help us learn more about whether people with a personal and/or family history of colorectal cancer and other cancers follow cancer screening recommendations.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be eligible for enrollment if he/she is self-referred or physician-referred for genetic counseling at Memorial Sloan-Kettering Cancer Center's (MSKCC) Clinical Genetics Service due to a concern about increased risk for colon cancer or;
* An individual who presents for genetic counseling at MSKCC's Clinical Genetics Service after undergoing genetic testing at an outside institution with a documented mutation in any gene associated with Lynch Syndrome or;
* An individual who in the context of genetic counseling has received stricter colorectal and/or gynecologic screening recommendations than that of the general population regardless of genetic test results.
* DNA of patients who have been consented to protocol 93-102 ("Ascertainment of Peripheral Blood or Saliva Samples for Genetic Epidemiology Studies of Familial Cancers"), who meet the eligibility criteria listed above, will also be eligible for inclusion in this study.

Exclusion Criteria:

* Patients will be excluded from this study if: he/she has physical, cognitive or psychiatric conditions that interfere with ability to give meaningful informed consent; he/she cannot read, write or communicate in English; he/she is less than 18 years of age; he/she has received a diagnosis of FAP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking genetic counseling with or without genetic testing for colorectal cancer risk and/or suspected Lynch Syndrome will be recruited and offered enrollment during their first counseling visit at the Clinical Genetics Service at MSKCC
Sampling Method: Non-Probability Sample
Enrollment: 1530 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess adherence to comprehensive, multi-organ screening and risk-reducing behavior recommendations in patients with Lynch Syndrome. | conclusion of study

SECONDARY OUTCOMES:
To evaluate predictive factors for adherence to comprehensive, multi-organ screening and risk-reducing behavior recommendations. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Zsofia Stadler, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center Hauppauge (Consent Only), Hauppauge, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org